CLINICAL TRIAL: NCT04200677
Title: Influence of Electrode Positioning and Current Type on Muscle Fatigability, Force Generation, Perceived Discomfort and Neuromuscular Adaptations Induced by Neuromuscular Electric Stimulation: Implications on Rehabilitation
Brief Title: Influence of Electrode Positioning and Current Type on Fatigue, Force and Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Physical Therapist, Assistant Professor, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CAAE: 14734619.3.0000.8093
Record Dates: First submitted 2019-12-05; First posted 2019-12-16 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Electrical Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MCN1 (Experimental): Monophasic Current (100 Hz) with 1ms pulse width applied to the Tibial Nerve
  Interventions: Other: Monophasic Current (100 Hz) with 1ms pulse width applied to the Tibial Nerve
- BCN05 (Experimental): Biphasic current (100 Hz) with pulse width 0.5ms applied to the Tibial Nerve
  Interventions: Other: Biphasic current (100 Hz) with pulse width 0.5ms applied to the Tibial Nerve
- BCN1 (Experimental): Biphasic current (100 Hz) with 1ms pulse width applied to the Tibial Nerve
  Interventions: Other: Biphasic current (100 Hz) with 1ms pulse width applied to the Tibial Nerve
- BCN2 (Experimental): Biphasic current (100 Hz) with 2ms pulse width applied to the Tibial Nerve
  Interventions: Other: Biphasic current (100 Hz) with 2ms pulse width applied to the Tibial Nerve
- MCM1 (Experimental): Monophasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly
  Interventions: Other: Monophasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly
- BCM05 (Experimental): Biphasic current (100 Hz) with pulse width 0.5ms applied to the Triceps Surae muscle Belly
  Interventions: Other: Biphasic current (100 Hz) with pulse width 0.5ms applied to the Triceps Surae muscle Belly
- BCM1 (Experimental): Biphasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly
  Interventions: Other: Biphasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly
- BCM2 (Experimental): Biphasic current (100 Hz) with 2ms pulse width applied to the Triceps Surae Muscle Belly
  Interventions: Other: Biphasic current (100 Hz) with 2ms pulse width applied to the Triceps Surae Muscle Belly
- BC25 (Experimental): Biphasic current (25 Hz) with 0.5ms pulse width applied to the Triceps Surae Muscle Belly
  Interventions: Other: Biphasic current (25 Hz) with 0.5ms pulse width applied to the Triceps Surae Muscle Belly

INTERVENTIONS:
Other: Monophasic Current (100 Hz) with 1ms pulse width applied to the Tibial Nerve — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following NMES parameters: (Monophasic Current, 100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s)
  Arms: MCN1
Other: Biphasic current (100 Hz) with pulse width 0.5ms applied to the Tibial Nerve — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current, 100 Hz, pulse duration 0.5 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCN05
Other: Biphasic current (100 Hz) with 1ms pulse width applied to the Tibial Nerve — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current, 100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCN1
Other: Biphasic current (100 Hz) with 2ms pulse width applied to the Tibial Nerve — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current, 100 Hz, pulse duration 2 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCN2
Other: Monophasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Monophasic current, 100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s)
  Arms: MCM1
Other: Biphasic current (100 Hz) with pulse width 0.5ms applied to the Triceps Surae muscle Belly — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current, 100 Hz, pulse duration 0.5 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCM05
Other: Biphasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current , 100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCM1
Other: Biphasic current (100 Hz) with 2ms pulse width applied to the Triceps Surae Muscle Belly — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current , 100 Hz, pulse duration 2 ms, Ton: 6 s, Toff: 18 s)
  Arms: BCM2
Other: Biphasic current (25 Hz) with 0.5ms pulse width applied to the Triceps Surae Muscle Belly — The participants will perform 36 contractions evoked by neuromuscular electrical stimulation with the following current parameters: (Biphasic current, 25 Hz, pulse duration 0.5 ms, Ton: 6 s, Toff: 18 s)
  Arms: BC25

SUMMARY:
Introduction: Neuromuscular electrical stimulation (NMES) has the purpose of generating muscle contractions to minimize muscular atrophy and to improve neuromuscular performance. NMES has been performed using monophasic or biphasic currents, applied over a nerve trunk or muscle belly, and both can generate contractions by the peripheral and central nervous system. Pulse width (wide or narrow) is an essential parameter for NMES. Although NMES studies using wide pulses have been performed with monophasic currents, it is known that this current induces discomfort during NMES. Therefore, it is necessary to analyze if biphasic currents have the same effect as monophasic currents using the same parameters.

Objectives:

To compare the effects of NMES with narrow and wide pulse widths associated with monophasic and biphasic currents, applied over a tibial nerve and triceps surae muscles in healthy individuals in terms of muscle fatigue, central and peripheral contribution, voluntary and evoked force and sensory discomfort.

Methods:

A crossover, experimental controlled and randomized study will be developed with healthy male and female (age: 18-45 years). The following dependent variables will be: amplitude of H-reflex and M-wave (single and double pulses), voluntary and evoked triceps surae muscles torque, fatigability (force time integral), perceived discomfort and neuromuscular adaptations. The independent variables will be related to current phase, pulse width and location of electrical stimulation electrodes. There will be a familiarization session followed by 9 sessions with 7 rest days between them (10 weeks). Data will be reported as mean and standard deviation (± SD). Parametric tests will be used for the normally distributed data (Shapiro-Wilk test) that show homogeneous variations (Levene test). A repeated measure mixed-model ANOVA will be performed and, in the case of major effects or significant interactions, the Tukey post-hoc test will be applied. In addition, the power and size of the effect (reported as partial eta square, partial η2) will be calculated. The significance threshold will be set at p <0.05 for all procedures.

Expected results: Biphasic currents will be more comfortable and will generate less muscle fatigue when compared to monophasic currents. There will be less fatigue and greater central contribution when wider pulse currents will be applied over a nerve trunk concerning the application with a wide pulse over a muscle belly.

DETAILED DESCRIPTION:
This is a randomized controlled trial, a crossover study, with healthy male and female participants. The procedures will take place in 10 distinct visits for a 7-day interval.

The following visit in the lab will be:

* Familiarization session.
* Monophasic Current (100 Hz) with 1ms pulse width applied to the Tibial Nerve;
* Biphasic current (100 Hz) with pulse width 0.5ms applied to the Tibial Nerve;
* Biphasic current (100 Hz) with 1ms pulse width applied to the Tibial Nerve;
* Biphasic current (100 Hz) with 2ms pulse width applied to the Tibial Nerve;
* Monophasic (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly;
* Biphasic current (100 Hz) with pulse width 0.5ms applied to the Triceps Surae muscle Belly;
* Biphasic current (100 Hz) with 1ms pulse width applied to the Triceps Surae Muscle Belly;
* Biphasic current (100 Hz) with 2ms pulse width applied to the Triceps Surae Muscle Belly;
* Biphasic current (25 Hz) with 0.5ms pulse width applied to the Triceps Surae Muscle Belly.

The dependent variables will be:

* Muscle fatigability;
* Central and peripheral contribution (with H-reflex and M-wave amplitude analysis);
* Maximum voluntary isometric contraction;
* Force production for plantar flexion evoked by NMES;
* Perceived discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Classified as physically active according to the INTERNATIONAL QUESTIONNAIRE OF PHYSICAL ACTIVITY;
* To practice only recreational physical activity;
* Be at least 3 months without practicing strength training.

Exclusion Criteria:

* Present some type of skeletal muscle dysfunction that may interfere with the tests;
* NMES intolerance in the triceps surae muscle belly or tibial nerve;
* Use of analgesics, antidepressants, tranquilizers or other centrally acting agents;
* Cardiovascular or peripheral vascular problems, chronic diseases, neurological or muscular disorders that may hinder the complete execution of the study design by the volunteer.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle Fatigue | Change from baseline to the end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Muscle Fatigue will be assessed by Force time integral (area under the force trace), after neuromuscular electrical stimulation protocol.
Muscle Force | Change from baseline to the end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Muscle force will be assessed by muscle force changes, based on the torque generated pre and post neuromuscular electrical stimulation protocol.
Change from Baseline Central contribution (H reflex amplitude) after 15 minutes session of NMES | Change from baseline to the end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Central contribution will be measured before and after 15 minutes (36 contractions) of electrical stimulation in the session.
Change from Baseline Peripheral contribution (M wave amplitude) after 15 minutes session of NMES | Change from baseline to the end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Peripheral contribution will be measured before and after acute session 15 minutes (36 contractions) of electrical stimulation in the session.
Change from Baseline Evoked Torque after 15 minutes session of electrical stimulation | Change from baseline to the end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Evoked Torque will be measured before and after acute session 15 minutes (36 contractions) of electrical stimulation in the session.
Discomfort | At the beginning, middle and end of thirty-six contractions evoked by electrical stimulation (1 per week, total of 9 sessions). This outcome will be measured up to 9 weeks. Data will be reported through study completion (4 years).
  Discomfort sensory will be evaluated by Visual Analogic Scale during and after the evoked torque measurement with NMES. The Visual Analogic Scale assess pain by rating the subjective perceived discomfort of the subject from 0 (no perceived discomfort) to 10 (the most perceived discomfort)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - University of Brasília, Brasília, Federal District
  - Faculty of Physical Education, Brasília, Federal District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ward AR, Robertson VJ. The variation in fatigue rate with frequency using kHz frequency alternating current. Med Eng Phys. 2000 Nov;22(9):637-46. doi: 10.1016/s1350-4533(00)00085-0. PMID 11259932
- [Background] Aldayel A, Jubeau M, McGuigan M, Nosaka K. Comparison between alternating and pulsed current electrical muscle stimulation for muscle and systemic acute responses. J Appl Physiol (1985). 2010 Sep;109(3):735-44. doi: 10.1152/japplphysiol.00189.2010. Epub 2010 Jul 1. PMID 20595542
- [Background] Ward AR, Lucas-Toumbourou S, McCarthy B. A comparison of the analgesic efficacy of medium-frequency alternating current and TENS. Physiotherapy. 2009 Dec;95(4):280-8. doi: 10.1016/j.physio.2009.06.005. Epub 2009 Sep 2. PMID 19892092
- [Background] Selkowitz DM, Rossman EG, Fitzpatrick S. Effect of burst-modulated alternating current carrier frequency on current amplitude required to produce maximally tolerated electrically stimulated quadriceps femoris knee extension torque. Am J Phys Med Rehabil. 2009 Dec;88(12):973-8. doi: 10.1097/PHM.0b013e3181c1eda5. PMID 19935181
- [Background] Ward AR, Shkuratova N. Russian electrical stimulation: the early experiments. Phys Ther. 2002 Oct;82(10):1019-30. PMID 12350217
- [Background] Bergquist AJ, Clair JM, Collins DF. Motor unit recruitment when neuromuscular electrical stimulation is applied over a nerve trunk compared with a muscle belly: triceps surae. J Appl Physiol (1985). 2011 Mar;110(3):627-37. doi: 10.1152/japplphysiol.01103.2010. Epub 2010 Dec 23. PMID 21183628
- [Background] Collins DF. Central contributions to contractions evoked by tetanic neuromuscular electrical stimulation. Exerc Sport Sci Rev. 2007 Jul;35(3):102-9. doi: 10.1097/jes.0b013e3180a0321b. PMID 17620928
- [Background] Martin A, Grospretre S, Vilmen C, Guye M, Mattei JP, LE Fur Y, Bendahan D, Gondin J. The Etiology of Muscle Fatigue Differs between Two Electrical Stimulation Protocols. Med Sci Sports Exerc. 2016 Aug;48(8):1474-84. doi: 10.1249/MSS.0000000000000930. PMID 27031743
- [Background] Neyroud D, Dodd D, Gondin J, Maffiuletti NA, Kayser B, Place N. Wide-pulse-high-frequency neuromuscular stimulation of triceps surae induces greater muscle fatigue compared with conventional stimulation. J Appl Physiol (1985). 2014 May 15;116(10):1281-9. doi: 10.1152/japplphysiol.01015.2013. Epub 2014 Mar 27. PMID 24674861
- [Background] Regina Dias Da Silva S, Neyroud D, Maffiuletti NA, Gondin J, Place N. Twitch potentiation induced by two different modalities of neuromuscular electrical stimulation: implications for motor unit recruitment. Muscle Nerve. 2015 Mar;51(3):412-8. doi: 10.1002/mus.24315. Epub 2015 Jan 5. PMID 24917022
- [Background] Wegrzyk J, Foure A, Le Fur Y, Maffiuletti NA, Vilmen C, Guye M, Mattei JP, Place N, Bendahan D, Gondin J. Responders to Wide-Pulse, High-Frequency Neuromuscular Electrical Stimulation Show Reduced Metabolic Demand: A 31P-MRS Study in Humans. PLoS One. 2015 Nov 30;10(11):e0143972. doi: 10.1371/journal.pone.0143972. eCollection 2015. PMID 26619330
- [Background] Wegrzyk J, Foure A, Vilmen C, Ghattas B, Maffiuletti NA, Mattei JP, Place N, Bendahan D, Gondin J. Extra Forces induced by wide-pulse, high-frequency electrical stimulation: Occurrence, magnitude, variability and underlying mechanisms. Clin Neurophysiol. 2015 Jul;126(7):1400-12. doi: 10.1016/j.clinph.2014.10.001. Epub 2014 Oct 13. PMID 25454283
- [Background] Kiernan MC, Lin CS, Burke D. Differences in activity-dependent hyperpolarization in human sensory and motor axons. J Physiol. 2004 Jul 1;558(Pt 1):341-9. doi: 10.1113/jphysiol.2004.063966. Epub 2004 May 14. PMID 15146048
- [Background] Kiernan MC, Mogyoros I, Burke D. Differences in the recovery of excitability in sensory and motor axons of human median nerve. Brain. 1996 Aug;119 ( Pt 4):1099-105. doi: 10.1093/brain/119.4.1099. PMID 8813274
- [Background] Alexandre F, Derosiere G, Papaiordanidou M, Billot M, Varray A. Cortical motor output decreases after neuromuscular fatigue induced by electrical stimulation of the plantar flexor muscles. Acta Physiol (Oxf). 2015 May;214(1):124-34. doi: 10.1111/apha.12478. Epub 2015 Mar 18. PMID 25740017
- [Background] Dreibati B, Lavet C, Pinti A, Poumarat G. Influence of electrical stimulation frequency on skeletal muscle force and fatigue. Ann Phys Rehabil Med. 2010 May;53(4):266-71, 271-7. doi: 10.1016/j.rehab.2010.03.004. Epub 2010 Apr 1. English, French. PMID 20430713
- [Background] Jubeau M, Zory R, Gondin J, Martin A, Maffiuletti NA. Effect of electrostimulation training-detraining on neuromuscular fatigue mechanisms. Neurosci Lett. 2007 Aug 31;424(1):41-6. doi: 10.1016/j.neulet.2007.07.018. Epub 2007 Aug 1. PMID 17709192
- [Background] Hwang IS, Huang CY, Wu PS, Chen YC, Wang CH. Assessment of H reflex sensitivity with M wave alternation consequent to fatiguing contractions. Int J Neurosci. 2008 Sep;118(9):1317-30. doi: 10.1080/00207450802055606. PMID 18698513
- [Background] Boerio D, Jubeau M, Zory R, Maffiuletti NA. Central and peripheral fatigue after electrostimulation-induced resistance exercise. Med Sci Sports Exerc. 2005 Jun;37(6):973-8. PMID 15947722
- [Background] Foure A, Nosaka K, Wegrzyk J, Duhamel G, Le Troter A, Boudinet H, Mattei JP, Vilmen C, Jubeau M, Bendahan D, Gondin J. Time course of central and peripheral alterations after isometric neuromuscular electrical stimulation-induced muscle damage. PLoS One. 2014 Sep 12;9(9):e107298. doi: 10.1371/journal.pone.0107298. eCollection 2014. PMID 25215511